CLINICAL TRIAL: NCT01383980
Title: A Randomized Trial of Continuous Versus Interrupted Enteral Feeding in Critically Ill Surgical Patients Requiring Mechanical Ventilation
Brief Title: Trial of Continuous Versus Interrupted Feeding for Intubated Intensive Care Unit Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Laszlo Kiraly, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 00006259
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Malnutrition
Keywords: Enteral Nutrition; Enteral Feeding; nasogastric tubes; gastrostomy tubes; jejunostomy tubes
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Intervention Model Description: Subjects are randomized to remain NPO at midnight prior to surgery or to continue to receive tube feeding up until surgery time.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Tube feeds are held night prior to elective surgery (standard of care)
- Continuous Feeding (Experimental): Tube feeds are continued up until surgery. Subjects with a nasogastric tube will have their stomach contents emptied prior to surgery.
  Interventions: Dietary Supplement: Continuous Tube Feedings

INTERVENTIONS:
Dietary Supplement: Continuous Tube Feedings — Tube feeds continued up until elective surgery.
  Arms: Continuous Feeding

SUMMARY:
Surgical patients fed up until the point of surgery will have safe delivery of more calories compared to a group whose feeding is held at midnight prior to surgery.

DETAILED DESCRIPTION:
Nutrition is essential for healing and recovery from illness. Tube feeds are the standard care for patients with prolonged stays in the intensive care unit (ICU) who cannot eat food on their own. Tube feeding means that a tube has been placed in a patient's stomach or small intestine to provide nutrition.

When a patient is scheduled for an elective surgery, he/she usually has nothing to eat after midnight prior to the operation. A fasting period before surgery is done to avoid possible side effects during the placement of a breathing tube. Having an empty stomach is thought to decrease the chances of vomiting or aspiration while a breathing tube is placed. (Aspiration occurs when a substance, such as food provided by a tube feed, enters the airway.) However, some patients already have a breathing tube in place. The investigators do not know which is better for patients who already have a breathing tube in place: continuing feedings up until surgery or stopping them the night before.

The investigators hypothesize intubated surgical patients randomized to a protocol of feeding up until the point of surgery will have the safe delivery of more calories as compared to a group whose feeding is held at midnight prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Intubated with planned visit to the OR
* Admitted to an ICU at OHSU
* Receiving enteral nutrition or plan to start enteral nutrition

Exclusion Criteria:

* Age less than 18 years
* Unable to obtain consent from patient or ARR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Total calories delivered | Daily for length of stay (LOS). LOS defined as time from admission to discharge. LOS estimated to average three (3) weeks per participant.
  The total number of calories subject consume while receiving tube feeding.

SECONDARY OUTCOMES:
Laboratory values | Daily for length of stay (LOS). LOS defined as time from admission to discharge. LOS estimated to average three (3) weeks per participant.
  Laboratory values of interest include: CBC, liver function tests, basic metabolic panel, magnesium, phosphate, alubmin, prealubumin, c-reactive protein, and arterial blood gas.
Weight change | Daily for length of stay (LOS). LOS defined as time from admission to discharge. LOS estimated to average three (3) weeks per participant.
  The change of weight during hospital admission.
number of infections and aspiration events | From date of randomization until the date of documented complication. Subjects will be followed until discharge in case of multiple complications. Date of discharge is estimated to be three (3) weeks post-admission on average.
  Number of infections or aspiration events during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Laszlo Kiraly, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University (OHSU), Portland, Oregon, United States

REFERENCES:
- [Background] Braunschweig CL, Levy P, Sheean PM, Wang X. Enteral compared with parenteral nutrition: a meta-analysis. Am J Clin Nutr. 2001 Oct;74(4):534-42. doi: 10.1093/ajcn/74.4.534. PMID 11566654
- [Background] Kudsk KA, Croce MA, Fabian TC, Minard G, Tolley EA, Poret HA, Kuhl MR, Brown RO. Enteral versus parenteral feeding. Effects on septic morbidity after blunt and penetrating abdominal trauma. Ann Surg. 1992 May;215(5):503-11; discussion 511-3. doi: 10.1097/00000658-199205000-00013. PMID 1616387
- [Background] Kalfarentzos F, Kehagias J, Mead N, Kokkinis K, Gogos CA. Enteral nutrition is superior to parenteral nutrition in severe acute pancreatitis: results of a randomized prospective trial. Br J Surg. 1997 Dec;84(12):1665-9. PMID 9448611
- [Background] McClave SA, Martindale RG, Vanek VW, McCarthy M, Roberts P, Taylor B, Ochoa JB, Napolitano L, Cresci G; A.S.P.E.N. Board of Directors; American College of Critical Care Medicine; Society of Critical Care Medicine. Guidelines for the Provision and Assessment of Nutrition Support Therapy in the Adult Critically Ill Patient: Society of Critical Care Medicine (SCCM) and American Society for Parenteral and Enteral Nutrition (A.S.P.E.N.). JPEN J Parenter Enteral Nutr. 2009 May-Jun;33(3):277-316. doi: 10.1177/0148607109335234. No abstract available. PMID 19398613
- [Background] Jenkins ME, Gottschlich MM, Warden GD. Enteral feeding during operative procedures in thermal injuries. J Burn Care Rehabil. 1994 Mar-Apr;15(2):199-205. doi: 10.1097/00004630-199403000-00019. PMID 8195265
- [Background] Pousman RM, Pepper C, Pandharipande P, Ayers GD, Mills B, Diaz J, Collier B, Miller R, Jensen G. Feasibility of implementing a reduced fasting protocol for critically ill trauma patients undergoing operative and nonoperative procedures. JPEN J Parenter Enteral Nutr. 2009 Mar-Apr;33(2):176-80. doi: 10.1177/0148607108327527. PMID 19251911